CLINICAL TRIAL: NCT04679337
Title: Changes in Renal Tissue Oxygen Saturation and Its Relationship With Central Venous and Cerebral Oxygen Saturation During Off-pump Coronary Artery Bypass Graft Surgery
Brief Title: Renal Oxygen Saturation During Off-pump Coronary Artery Bypass Graft Surgery
Acronym: OPCAB
Status: Completed | Type: Observational
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Professor, Yeungnam University College of Medicine
Other Study IDs: YUMC-2020-11-035
Record Dates: First submitted 2020-12-08; First posted 2020-12-22 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Oximetry; Coronary Artery Bypass, Off-Pump
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate changes in renal oxygen saturation (rrSO2) and its relationship with central venous oxygen saturation (cvSO2), cerebral cortical oxygen saturation (rcSO2), and hemodynamic parameters while displacing the heart for each coronary anastomosis in 19-80 year old adult patients receiving off-pump coronary artery bypass graft surgery (OPCAB) under general anesthesia.

DETAILED DESCRIPTION:
In the current clinical trial, systemic perfusion and oxygenation through hemodynamic variables such as cardiac index and mean arterial pressure, and central venous oxygen saturation (cvSO2) are monitored during surgery. However, it has not been studied whether the hemodynamic parameters and systemic oxygen saturation adequately reflect the perfusion and oxygen saturation of the kidney. Although there are various new serum biomarkers that are known to reflect renal function or damage, they are not real-time monitoring of renal function because they take time and cost to collect and analyze.

Near-infrared spectroscopy (NIRS) measures the distribution of oxygenated hemoglobin and deoxygenated hemoglobin in tissues by sending two different near-infrared wavelengths (730 and 810 nm) from the sensor. It is a device that can continuously monitor the oxygen supply-demand balance to a specific region non-invasively. NIRS is mainly used to measure the oxygen demand-supply balance of the cerebral tissue by attaching a sensor to the forehead in the surgical patient. Since it is known to be closely related to the reduction of cerebral oxygen saturation during surgery and the occurrence of postoperative cognitive dysfunction, it is used as an indispensable monitoring device to prevent neurological complications in heart surgery patients. Recently, with technological advances, it has become possible to measure oxygen saturation by attaching sensors to various body tissues other than the brain. When monitored with an NIRS sensor attached to the kidney, the relationship between renal oxygen saturation reduction and postoperative acute kidney injury (AKI) in children and adult patients undergoing heart surgery was reported. However, so far, the effects of systemic hemodynamic and oxygen saturation changes during the displacement of heart for coronary anastomosis during OPCAB on the oxygen saturation in the cerebral cortex and kidney, have not been studied. In addition, it is not known whether the cerebral cortical oxygen saturation (rcSO2), which is commonly used in heart surgery, can reflect the renal oxygen saturation (rrSO2).

The purpose of this study is to evaluate changes in renal oxygen saturation (rrSO2) and its relationship with central venous oxygen saturation (cvSO2), cerebral cortical oxygen saturation (rcSO2), and hemodynamic parameters while displacing the heart for each coronary anastomosis in 19-80 year old adult patients receiving off-pump coronary artery bypass graft surgery (OPCAB) under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of coronary artery obstructive disease
* undergoing off-pump coronary artery bypass graft surgery

Exclusion Criteria:

* renal artery stenosis
* Hyperbilirubinemia (total bilirubin> 1.2 mg/dl)
* Kidney disease (serum creatinine 1.5 mg/dl) or chronic kidney failure
* Carotid artery stenosis (> 60%)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients between 19 and 80 years old undergoing off-pump coronary artery bypass graft surgery due to coronary artery ostructive disease
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
rrSO2 and cvSO2 | up tp 30 days after surgery
  Correlation between renal oxygen saturation and central venous oxygen saturation

SECONDARY OUTCOMES:
rrSO2 and rcSO2 | up to 30 days after surgery
  Correlation between renal oxygen saturation and cerebral oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Medical Center, Daegu, South Korea